CLINICAL TRIAL: NCT01375309
Title: Effect of Bifidobacterium Bifidum Supplementation on Morbidity of Very Low Birth Weight Infants
Brief Title: Bifidobacterium Supplementation for Very Low Birth Weight Infants
Acronym: Bifido(RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Women's Medical University (Other)
Responsible Party: Principal Investigator, Satoshi Kusuda, Professor of Neonatology, Tokyo Women's Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1675; UMIN000002543 (Other: University hospital Medical Information Network)
Record Dates: First submitted 2011-06-06; First posted 2011-06-17 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Preterm Infants
Keywords: probiotics; preterm infants; enteral feeding; Bifidobacterium on enteral feeding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Bifidobacterium bifidum
  Interventions: Dietary Supplement: Bifidobacterium bifidum supplementation
- Placebo (Placebo Comparator): Dextrin without Bifidobacterium bifidum
  Interventions: Dietary Supplement: Placebo contains dextrin

INTERVENTIONS:
Dietary Supplement: Bifidobacterium bifidum supplementation — Bifidobacterium bifidum supplementation wiht approximately 2.5*10to9th bacteria per day
  Other Names: Bifidobacterium bifidum OLB6378
  Arms: Active
Dietary Supplement: Placebo contains dextrin — 0.5 of dextrin
  Arms: Placebo

SUMMARY:
Probiotic supplementation to preterm infants have been reported to be beneficial in neonatal intensive care unit (NICU). Our pilot study also showed accelerated feeding in preterm infants who received Bifidobacterium bifidum early after birth. In order to evaluate these beneficial effects of Bifidobacterium bifidum, a prospective randomized control study is conducted. The hypothesis of the study is that Bifidobacterium bifidum supplementation to preterm infants improve enteral feeding and growth in very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants with birth weight less than 1500g

Exclusion Criteria:

* Sever bacteremia
* Congenital anomaly
* Not suitable for the trial defined by an attending neonatologist

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postnatal day when enteral feeding exceeded at 100ml/kg/day | From birth untill the date of enteral feeding first exceeded at 100ml/kg/day or date of death from any cause, whichever came first, assesed up to 27 days after birth
  Death or unsuccessful of establishing enteral feeding exceeded at 100ml/kg/day before day 28 of age is considered failure to reach primary endpoint.

SECONDARY OUTCOMES:
standard deviation(SD) scores of bodyweight(BW) and head circumference(HC) | For the duration of NICU stay, an expected average of 3 months
  BW gain/day, SD scores of BW and HC at discharge from NICU
Necrotizing enterocolitis or sepsis | For the duration of NICU stay, an expected average of 3 months
  The incidences of necrtizing enterocolitis or sepsis during the stay in NICU
Intestinal flora | For the duration of NICU stay, an expected average of 3 months
  Intestinal flora during the stay in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Kusuda, MD, Principal Investigator — Tokyo Women's Medical University
Locations (1):
- Tokyo Women's Medical Unversity, Shinjuku, Tokyo, Japan

REFERENCES:
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD005496. doi: 10.1002/14651858.CD005496.pub6. PMID 37493095
- [Derived] Sharif S, Meader N, Oddie SJ, Rojas-Reyes MX, McGuire W. Probiotics to prevent necrotising enterocolitis in very preterm or very low birth weight infants. Cochrane Database Syst Rev. 2020 Oct 15;10(10):CD005496. doi: 10.1002/14651858.CD005496.pub5. PMID 33058137